CLINICAL TRIAL: NCT05436964
Title: Effect of Intraoperative Dexmedetomidine on Postoperative Delirium in Elderly Patients Undergoing Major Abdominal Surgery: a Randomized Controlled Study
Brief Title: Effect of Intraoperative Dexmedetomidine on Postoperative Delirium in Elderly Patients Undergoing Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Hao Li, Associate professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChinesePLAGH301
Record Dates: First submitted 2022-06-26; First posted 2022-06-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2023-09

CONDITIONS: Delirium in Old Age
Keywords: dexmedetomidine
MeSH Terms: interventions — Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Use 250 ml of saline as placebo group.
  Interventions: Other: saline
- Experimental group (Experimental): Use dexmedetomidine as experimental group
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Other: saline — Patients in the experimental group were given a loading dose of 0.6 μg/kg of saline intravenously after 10 minutes of intubation, followed by a continuous infusion at a rate of 0.4 μg/kg/h until 30 min before the end of the surgery.continuous infusion at a rate of 0.4 μg/kg/h until 30 min before the end of the surgery.
  Arms: Placebo group
Drug: Dexmedetomidine — Patients in the experimental group were given a loading dose of 0.6 μg/kg of dexmedetomidine intravenously after 10 minutes of intubation, followed by a continuous infusion at a rate of 0.4 μg/kg/h until 30 min before the end of the surgery.
  Arms: Experimental group

SUMMARY:
To observe the effect of intraoperative dexmedetomidine on the incidence of postoperative delirium, postoperative analgesic drug requirements and pain scores in elderly patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled trial. Three hundred patients undergoing elective major abdominal surgery were randomized to the intervention and control groups. Patients in the intervention group were given a loading dose of 0.6 μg/kg of dexmedetomidine by intravenous infusion within 10 minutes after intubation, followed by a continuous infusion at a rate of 0.4 μg/kg/h until 30 min before the end of the procedure; patients in the control group were given an equal volume of saline. Data were collected at 1-5 days and 1 month postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old
* Patients undergoing elective major abdominal surgery
* Written informed consent was obtained

Exclusion Criteria:

* Patients with severe preoperative cognitive impairment (MMSE ≤ 20) who are unable to undergo a follow-up evaluation.
* Patients with history of psychiatric or neurological disorders.
* Patients with body mass index ≤ 18 or ≥ 30
* Patients with severe bradycardia (heart rate less than 40 beats per minute)
* Patients with pathological sinus node syndrome or grade 2 or greater AV block
* Patients with severe hepatic or renal insufficiency.
* Patients with severe hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 268 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Participants will be followed for the duration of hospital stay, an expected average of 5 days.Evaluations are conducted twice a day.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Li, Principal Investigator — Chinese PLA General Hospital
Locations (3):
- China (3):
  - Beijing Tiantan Hospital,Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - Central theater General Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No